CLINICAL TRIAL: NCT02495701
Title: Complications Related to Arthroscopic Surgery of the Hip - a Prospective Cohort Study
Status: Terminated | Type: Observational
Why Stopped: main outcome could not be ekstracted from database
Sponsor: University of Aarhus (Other)
Collaborators: Horsens Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 1-16-02-260-15
Record Dates: First submitted 2015-06-01; First posted 2015-07-13 (Estimated); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Hip Pathology; Femoracetabular Impingement
MeSH Terms: conditions — Femoracetabular Impingement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients: Patients having Hip arthroscopic surgery
  Interventions: Procedure: Hip arthroscopic surgery

INTERVENTIONS:
Procedure: Hip arthroscopic surgery — Hip arthroscopic surgery

SUMMARY:
Arthroscopic hip surgery is performed with traction on the leg to allow the surgeon to perform the surgical procedure. A retrospective study has described neuropraxia, ankle joint pain and a skin burn after surgery (1). Moreover, it has been described that surgeons performing the procedure have a learning curve related to the number of complications described postoperatively. At the investigators' institution, hip arthroscopies have been performed since 2010 and the 3 surgeons have 4-12 years of experience. During the past years, changes have been made to secure the best possible comfort for the patient during the arthroscopic procedure. Hence, there is a rationale for investigating complications after hip arthroscopy in a setting that is less affected by the surgeon's learning curve and with the patient comfort in focus.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing hip arthroscopic surgery at Horsens Hospital, Denmark, during one year.

Exclusion Criteria:

* Non

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing hip arthroscopic surgery at Horsens Hospital, Denmark
Sampling Method: Non-Probability Sample
Enrollment: 220 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2022-12-15 (Actual)

PRIMARY OUTCOMES:
Visual analog scale-pain of the knee | Three months after surgery
Visual analog scale-pain of the ankle | Three months after surgery
Number of patients reporting numbness | Three months after surgery
Number of adverse events | From surgery to one year after surgery
  Infections, deep vein thrombosis, caput femoris necrosis, fracture, nerve injuries

SECONDARY OUTCOMES:
Visual analog scale-pain of the hip/groin at rest | Two weeks after surgery
Visual analog scale-pain of the hip/groin at rest | Three months after surgery
Visual analog scale-pain of the hip/groin after activities | Two weeks after surgery
Visual analog scale-pain of the hip/groin after activities | Three months after surgery
Visual analog scale-pain of the knee | Two weeks after surgery
Visual analog scale-pain of the ankle | Two weeks after surgery
Number of patients reporting numbness | From surgery to two weeks after surgery
Number of patients reporting sexual dysfunction | From surgery to three months after surgery
Number of patients and areas where patients report pain (Pain drawings) | Two weeks after surgery
Number of patients and areas where patients report pain (Pain drawings) | Three months after surgery
Number of patients reporting superficial skin abrasion | From surgery to two weeks after surgery
Visual analog scale-pain of the back | Two weeks after surgery
Visual analog scale-pain of the back | Three months after surgery

OTHER OUTCOMES:
Patient reported symptoms from the hip | From surgery to one year after surgery
  Patients are requested to report if they hear clicks or other sounds from their hip
Treatments of the hip | From surgery to one year after surgery
  Patients are asked if they have had further surgery, injections etc. in their operated hip during the past year
State of the contralateral hip | From surgery to one year after surgery
  Patients are asked if they have had surgery or injections of their contralateral hip

CONTACTS AND LOCATIONS:
Locations (1):
- Horsens Regional Hospital, Horsens, Denmark

REFERENCES:
- [Background] Park MS, Yoon SJ, Kim YJ, Chung WC. Hip arthroscopy for femoroacetabular impingement: the changing nature and severity of associated complications over time. Arthroscopy. 2014 Aug;30(8):957-63. doi: 10.1016/j.arthro.2014.03.017. Epub 2014 May 14. PMID 24835839